CLINICAL TRIAL: NCT04150263
Title: Dislocated Intraocular Lenses: Effect of Modification of Surgical Repositioning and Capsular Fibrosis Impact on Position of IOL After Fixation Surgery in a Randomized Trial
Brief Title: Modification of Scleral Suture Fixation of Dislocated IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Erik Eye Hospital (Other)
Collaborators: Umeå University (Other)
Responsible Party: Principal Investigator, Laura Armonaite, Principal investigator, St. Erik Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/1838 - 31/2
Record Dates: First submitted 2019-10-29; First posted 2019-11-04 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Dislocated Intraocular Lens
Keywords: intraocular lens, dislocation
MeSH Terms: conditions — Joint Dislocations | interventions — Lenses, Intraocular

STUDY DESIGN:
Intervention Model Description: 1 arm included 56 patients, the other arm included 61 patients. Sixty controls with ordinary pseudophakia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional IOL repositioning (Other): Intraocular lens (IOL) ab externo scleral suture fixation
  Interventions: Procedure: Intraocular lens (IOL) ab externo scleral suture fixation
- Modification of traditional IOL repositioning (Other): Modified intraocular lens (IOL) ab externo scleral suture fixation
  Interventions: Procedure: Modified IOL ab externo scleral suture fixation

INTERVENTIONS:
Procedure: Intraocular lens (IOL) ab externo scleral suture fixation — traditional IOL scleral suture fixation
  Arms: Traditional IOL repositioning
Procedure: Modified IOL ab externo scleral suture fixation — Modified IOL scleral suture fixation
  Arms: Modification of traditional IOL repositioning

SUMMARY:
A prospective randomized study on patients with late in the bag intraocular lens (IOL) dislocation after cataract surgery. Two surgical techniques of suturing of IOL to the sclera will be compared in the study. IOL position will be compared between those two groups, as well to a control group consisting of ordinary pseudophakia where only measurement of IOL position will be performed.

DETAILED DESCRIPTION:
In this prospective randomized study 60 patients will be included with late intraocular lens (IOL) dislocation and 60 patients in a control group with ordinary pseudophakia. Traditional surgery includes a capsular-IOL complex fixation to sclera by looping a prolene suture not only around haptics but also through capsular tissue. Such a suture may cut through the bag, which may result in a decentered IOL. A modification of "the traditional" method was created at S:t Eriks Eye Hospital in order to achieve better centration of the IOL. The study will evaluate the efficacy of these two methods. Additionally, the impact of fibrosis of capsular bag on IOL stability postoperatively will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients with in-the-bag dislocated IOL who agree to participate in the study
* Inclusion criteria for the control group: pseudophakic eyes 7-10 years after uneventful cataract surgery.

Exclusion Criteria:

* patients with dislocated IOL that is not visible in the pupillary plane
* IOL design not suitable for suturing using capsular bag
* patients who are not able to cooperate under measurements
* patients with Marfan syndrome and ectopia lentis
* exclusion criterion for the control group: other eye surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
IOL position | through study completion, an average of 1,5 years
  Measured at 3 time points: 1 month, 6 months and 1.5 years postoperatively, with anterior optical coherence tomography (OCT).
Capsular thickness | preoperatively or as soon as possible postoperatively
  Measured with OCT and photographed on slit-lamp examination.
Astigmatism | through study completion, an average of 1,5 years
  Measured with corneal topography, autorefractometer and keratometer. Corneal and IOL related astigmatism measured in diopters.Measured at 3 time points: 1 month, 6 months and 1.5 years postoperatively,

SECONDARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | through study completion, an average of 1,5 years
  Measure for visual function. Measured in logMAR. Measured preoperatively, 1 month, 6 months and 1.5 years postoperatively
Intraocular Pressure (IOP) | through study completion, an average of 1,5 years
  Measure for the pressure inside the eye measured with Goldman applanation tonometer and iCare, both in mmHg. Measured preoperatively, 1 month, 6 months and 1.5 years postoperatively
administration of IOL lowering therapy | through study completion, an average of 1,5 years
  number of patients who used IOL lowering therapy
Number of participants with postoperative complications | through study completion, an average of 1,5 year
  Number of patients with retinal detachment, macular edema and other.
Precision of the IOL position measurement with OCT | 1 month or any other postoperative control through study completion, an average of 1,5 year
  Measurements of IOL position with OCT will be done 3 times by the same investigator in both mydriatic and non-mydriatic pupil status.
inflammation in anterior chamber | through study completion, an average of 1,5 years
  Measured at 2 time points: 6 months and 1.5 years postoperatively, with laser flare meter.

CONTACTS AND LOCATIONS:
Locations (1):
- Laura Armonaite, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No